CLINICAL TRIAL: NCT05702567
Title: The Effectiveness of Transvaginal Radiofrequency and Pelvic Floor Muscle Training Compared to Pelvic Floor Muscle Training in Women With Stress Urinary Incontinence: a Double-blind Randomized Controlled Trial
Brief Title: The Effectiveness of Transvaginal Radiofrequency in Women With Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: José Casaña Granell (Other)
Collaborators: University of Alcalá. Physiotherapy in Women's Health (FPSM) Research Group. (Unknown)
Responsible Party: Sponsor-Investigator, José Casaña Granell, Director, Head of the Department of Physiotherapy (University of Valencia), Clinical Professor., University of Valencia
Organization: University of Valencia (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: UV-INV_ETICA-1104660
Record Dates: First submitted 2022-12-12; First posted 2023-01-27 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Urinary Incontinence,Stress; Pelvic Floor Disorders; Urinary Incontinence; Pelvic Floor Muscle Weakness
Keywords: Urinary loss; Pelvic floor dysfunctions; Women; Pelvic floor muscle training; Indiba Therapy; Physiotherapy
MeSH Terms: conditions — Urinary Incontinence, Stress; Pelvic Floor Disorders; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: The present study is a double-blind randomized clinical trial. Two groups are located, case group and placebo group.
  The total number of sessions will be 18 sessions per patient, divided into three sessions per week for a total of six weeks. These sessions last one hour, with a net treatment time of 40 minutes in the supine position.
  The vaginal probe is inserted into the cavity using a lubricant suitable for intracavitary use and RF, the device is turned on, while the RF is applied, pelvic floor contractions are performed guided by the physiotherapist 2 (Marta Martínez Colmenar) .
  The evaluations before and after the study will be carried out by the physiotherapist 1 (Yasmin Er Rabiai Boudallaa) who is blinded to group allocation. All participants will be assessed before, after six weeks and 6 months after the start of the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The INDIBA radiofrequency device is randomized in a total of 99 programs, and in order of arrival, a number is assigned to each patient in which the intervention of the number is unknown. Patients will always be treated with the same program number, throughout all sessions.
  The evaluations of the study will be carried out by the physiotherapist 1 (Yasmin Er Rabiai Boudallaa) who is blinded during the clinical trial.
  And by the physiotherapist 2 (Marta Martínez Colmenar), is the responsible for the treatment of patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RF + PFMT (Experimental): The participants recieve 18 sessions of radiofrequency (RF) and pelvic floor muscle training (PFMT), divided into three sessions per week for a total of six weeks, with a net treatment time of 40 minutes, each one.
  Interventions: Device: RF + PFMT
- PFMT (Placebo Comparator): The participants recieve 18 sessions of no radiofrequency (RF) and pelvic floor muscle training (PFMT), divided into three sessions per week for a total of six weeks, with a net treatment time of 40 minutes, each one. The RF device is started, but in this case, the program does not work or apply radiofrequency to the patients.
  Interventions: Other: PFMT + Placebo RF

INTERVENTIONS:
Device: RF + PFMT — During each session the patient is lying face up, with knees bent and feet resting on the stretcher.
  Then, the vaginal probe is introduced into the cavity using a lubricant suitable for intracavitary use and radiofrequency. The device is started at 15% intensity and adapting to a 10-point Likert scale, at point 3 or 4 of intensity.
  At the same time that the radiofrequency is applied, pelvic floor contractions are performed guided by the physiotherapist, and these contractions are three:
  * 10 fast contractions of one second each, with 10 seconds of rest.
  * 5 seconds of sustained contraction and 10 seconds of rest.
  * 10 seconds of contraction maintained with 10 seconds of rest.
  The contraction maintenance time will be adapted to what each woman can keep the pelvic floor contracted, with a view to the goal being to complete these exercises cyclically during the entire session.
  Other Names: INDIBA Activ CT9 SN: 19A150410
  Arms: RF + PFMT
Other: PFMT + Placebo RF — The intervention is exactly the same as the group RF + PFMT, unlike the non-functioning of the RF in the patients belonging to this group.
  The patient is lying face up, with knees bent and feet resting on the stretcher. Then, the vaginal probe is introduced into the cavity using a lubricant suitable for intracavitary use and radiofrequency, the device is started at 15% intensity, but in this case, the program does not work or apply radiofrequency to the patients.
  At the same time, that the radiofrequency's probe is applied, pelvic floor contractions are performed guided by the physiotherapist, and these contractions are the three named in the Radiofrequency + PFMT.
  The contraction maintenance time will be adapted to what each woman can keep the pelvic floor contracted, with a view to the goal being to complete these exercises cyclically during the entire session.
  Other Names: INDIBA Activ CT9 SN: 19A150410
  Arms: PFMT

SUMMARY:
The following clinical trial investigates the efficacy of transvaginal radiofrequency in the physiotherapy treatment of stress urinary incontinence (SUI). The treatment compares transvaginal radiofrequency with pelvic floor muscle training (PFMT) and PFMT alone.

The present study is a randomized controlled trial with double blinding (evaluator and patients).

The objective is to evaluate what radiofrequency can provide in the improving of the quality of life, symptoms and pelvic floor muscle strength of patients with SUI.

The reason for the combination with PFMT, is that it is the golden standard treatment in pelvic floor rehabilitation and SUI improvement.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is a health burden for more than 200 million people in the world. 34% of women over the age of 40 experience or have already experienced some significant experience with UI, thus affecting their health-related quality of life (QoHR).

SUI is endowed with a complex and multifactorial pathophysiology, generally involving the pelvic floor musculature and adjacent collagen-dependent tissues that help in support.

According to the literature, there are two clearly described mechanisms:

* The loss of urethral support, of the anterior vaginal wall, transforming into urethral hypermobility.
* Deficiency of urethral closure, such as rotational descent of the proximal part of the urethra, of the pubourethral ligament, with loss of internal urethral integrity.

The pelvic floor musculature plays an important role in helping the urethral support, during voluntary contraction. If the muscles are weak, urine loss is greater.

RF is an electrophysical and medical technique that generates tissue heating for therapeutic purposes. This technology uses electromagnetic RF fields with frequencies between 434 and 925 MHz, these forming part of the techniques classified as high frequency. The increases in temperature can reach 41.5ºC to 45ºC, according to some studies, and in another reaching 50ºC, acting at 6 and 8 cm3 depth, and generating biological effects on the skin and in the deeper layers.

It is known that RF promotes angiogenesis and increases local vascularization, stimulating collagen and elastin, resulting in changes in the helical structure of collagen, due to the denaturation and restructuring of its fibers. Changing the nature of connective tissues.

Investigators will make use of the non-ablative resistive RF mode, which does not have the capacity to section, but does have cell stimulation through superficial application on the skin, generating anti-inflammatory effects at the physiological level and collagen contraction, as an effect of short duration, and the stimulation of collagen synthesis or neocollagenesis thanks to the inflammation of the fibroblasts, to repair the damage present, as a long-lasting effect. Which would be interesting, because the pelvic floor is formed in its great majority by connective tissue and this would help to regenerate the tissue.

Treatment with this technology has not been sufficiently investigated in the intravaginal treatment of the pelvic floor. Previous studies lead to transurethral medical treatments that require local anesthesia, and the pathologies treated are the different types of urinary incontinence (stress, urgency, and mixed) and vaginal laxity. However, from the transvaginal approach the investigators found few studies.

ELIGIBILITY:
Inclusion Criteria:

* Women between 20 - 75 years
* Previously diagnosed SUI through assessment and questionnaires.
* PAD Test of 1h with > or = 1gr of urine loss.
* Urine losses in the last week.
* Nulliparous and multiparous.

Exclusion Criteria:

* Women > 75 years.
* Another type of urinary incontinence, urge or mixed.
* Difficulty urinating
* Hematuria
* Pregnancy
* Patients with any type of cancer or with a personal history of it.
* Previous surgeries for the treatment of SUI
* Gynecological surgeries (hysterectomy, containment mesh for different prolapses).
* Neurological and cognitive problems.
* Injury to the spinal cord, lower limbs or pelvis.
* Grade II, III or IV pelvic organ prolapse.
* Vaginal or urinary infection.
* Drugs:

  * Antimuscarinics (oxybutinin)
  * Toterodine
  * Trospium
  * Solifenacin
  * Darifenacin
  * Fesoterodine
  * Atropine
  * Anticholinergics
  * Antidepressants:
  * Duloxetine
  * Imipramine
  * Estrogens
  * Botulinum Toxin
  * Alpha-adrenergic agonists
  * Ephedrine
  * Pseudoephedrine
  * Antidiuretics (desmopressin)

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Changes in the ICIQ-SF scale before, after and six months after treatment in both groups. | Before treatment, six weeks of treatment, and 6 months assessments were required.
  ICIQ-SF: International Consultation on Incontinence Questionnaire, short form. The minimum score is 0, and the maximum is 21. Where 0 is the absence of urinary incontinence and everything valued above 0 is a symptom of urinary incontinence. The higher the value, the worse the incontinence.
The change of signs, symptoms and impact of pelvic floor dysfunction (PFDI-20) between reviews (before, after and at six months of treatment in both groups). | Before treatment, six weeks of treatment, and 6 months assessments were required.
  PFDI-20 : Pelvic Floor Distress Inventory Questionnaire - 20. It has 20 questions that are in turn divided into three symptomatic scales.
  The minimum value is 0, and the maximum is 300, which is the result of the sum of the total of the three subscales of 100 points of maximum value. This scale, the higher the value, the greater the pelvic floor dysfunction.
The change of signs, symptoms and impact of pelvic floor dysfunction (PFIQ-7) between reviews (before, after and at six months of treatment in both groups) | Before treatment, six weeks of treatment, and 6 months assessments were required.
  PFIQ-7 has 7 questions for each subscale, which are three in total. The minimum value is 0, and the maximum is 300, which is the result of the sum of the total of the three subscales of 100 points of maximum value. This scale, the higher the value, the greater the pelvic floor dysfunction.

SECONDARY OUTCOMES:
Changes in maximum and average strength of the pelvic floor before, after and six months after treatment in both groups. . | Before treatment, six weeks of treatment, and 6 months assessments were required.
  The maximum and average muscle strength is the value offered by the pelvimetry at the vaginal level, resulting from three submaximal contractions requested from the woman.
Changes in muscle tone before, after and six months after treatment in both groups. | Before treatment, six weeks of treatment, and 6 months assessments were required.
  Muscle tone is measured with a pelvimeter, which is inserted vaginally and the patient in the supine position and triple flexion of the lower limbs, relaxes and we take the base measurement, resulting from the subtraction of the result obtained minus 170mmHg of base.
Changes in sexual function (FSFI) before, after and six months after treatment in both groups. | Before treatment, six weeks of treatment, and 6 months assessments were required.
  FSFI: Female Sexual Function Index. The minimum value is 2, and the maximum is 36, which is the result of the sum of the results of each domain, which are 6 in total, with a maximum value of 6 points each. This scale the higher the value, the better sexual function.
  It consists of 19 questions, divided into subgroups according to the symptom to be studied: desire, arousal, lubrication, orgasm, satisfaction, and pain.
Check the level of physical activity measured with the GPAQ scale, in both groups, before, after and at six months. | Before treatment, six weeks of treatment, and 6 months assessments were required.
  GPAQ: global physical activity questionnaire. The GPAQ measures how many MET-min of physical activity is engaged during a typical week. The MET-min per week obtained from the GPAQ is a scale-type variable. Moderate- intensity physical activity corresponds to 4 MET/min, and vigorous-intensity physical activity corresponds to 8 MET/min.[6] During the calculation of weekly total MET-min, the durations of each type of physical activity are multiplied by these coefficients.
  The minimum value is 0 and the maximum is 3000 MET-min.
Changes in the Pad Test 1h before, after and six months after treatment in both groups. | Before treatment, six weeks of treatment, and 6 months assessments were required.
  Indications are given for one consecutive hour using a pad that will be given to the researcher, as well as a pad of the same model to weigh the difference obtained. The indications range from the intake of 500 ml of water, to various abdominal hyperpressure exercises.
Changes in Pelvic Muscle Excersice Self-Efficacy (Broome scale) before, after and six months after treatment in both groups. | Before treatment, six weeks of treatment, and 6 months assessments were required.
  Evaluates the perception and safety of patients in knowing how to contract the pelvic floor in different situations of daily life and their degree of confidence in them in the face of abdominal hyperpressure.
  The minimum value is 0 and the maximum is 100 in both subscales. The higher the value, the greater the awareness and confidence in the pelvic floor contractions.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Er Rabiai Boudallaa, Phd Student, Principal Investigator — University of Valencia (Spain)
Locations (1):
- Yasmin Er Rabiai Boudallaa, San Agustín del Guadalix, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buchsbaum GM, McConville J, Korni R, Duecy EE. Outcome of transvaginal radiofrequency for treatment of women with stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Mar;18(3):263-5. doi: 10.1007/s00192-006-0136-4. Epub 2006 Jun 21. PMID 16788852
- [Background] Lukban JC. Transurethral radiofrequency collagen denaturation for treatment of female stress urinary incontinence: a review of the literature and clinical recommendations. Obstet Gynecol Int. 2012;2012:384234. doi: 10.1155/2012/384234. Epub 2011 Oct 12. PMID 22007230
- [Background] KEGEL AH, POWELL TO. The physiologic treatment of urinary stress incontinence. J Urol. 1950 May;63(5):808-14. doi: 10.1016/S0022-5347(17)68832-3. No abstract available. PMID 15422687
- [Result] Kumaran B, Watson T. Thermal build-up, decay and retention responses to local therapeutic application of 448 kHz capacitive resistive monopolar radiofrequency: A prospective randomised crossover study in healthy adults. Int J Hyperthermia. 2015;31(8):883-95. doi: 10.3109/02656736.2015.1092172. Epub 2015 Nov 2. PMID 26524223
- [Result] Giombini A, Giovannini V, Di Cesare A, Pacetti P, Ichinoseki-Sekine N, Shiraishi M, Naito H, Maffulli N. Hyperthermia induced by microwave diathermy in the management of muscle and tendon injuries. Br Med Bull. 2007;83:379-96. doi: 10.1093/bmb/ldm020. PMID 17942453
- [Result] Smith WB, Melton W, Davies J. Midsubstance Tendinopathy, Percutaneous Techniques (Platelet-Rich Plasma, Extracorporeal Shock Wave Therapy, Prolotherapy, Radiofrequency Ablation). Clin Podiatr Med Surg. 2017 Apr;34(2):161-174. doi: 10.1016/j.cpm.2016.10.005. Epub 2017 Jan 18. PMID 28257672
- [Result] Lalji S, Lozanova P. Evaluation of the safety and efficacy of a monopolar nonablative radiofrequency device for the improvement of vulvo-vaginal laxity and urinary incontinence. J Cosmet Dermatol. 2017 Jun;16(2):230-234. doi: 10.1111/jocd.12348. Epub 2017 May 29. PMID 28556393
- [Result] Herman RM, Berho M, Murawski M, Nowakowski M, Rys J, Schwarz T, Wojtysiak D, Wexner SD. Defining the histopathological changes induced by nonablative radiofrequency treatment of faecal incontinence--a blinded assessment in an animal model. Colorectal Dis. 2015 May;17(5):433-40. doi: 10.1111/codi.12874. PMID 25524045
- [Result] Sodre DSM, Sodre PRS, Brasil C, Teles A, Doria M, Cafe LE, Lordelo P. New concept for treating urinary incontinence after radical prostatectomy with radiofrequency: phase 1 clinical trial. Lasers Med Sci. 2019 Dec;34(9):1865-1871. doi: 10.1007/s10103-019-02784-7. Epub 2019 Apr 15. PMID 30989457
- [Result] Caruth JC. Evaluation of the Safety and Efficacy of a Novel Radiofrequency Device for Vaginal Treatment. Surg Technol Int. 2018 Jun 1;32:145-149. PMID 29791707
- [Result] Kang D, Han J, Neuberger MM, Moy ML, Wallace SA, Alonso-Coello P, Dahm P. Transurethral radiofrequency collagen denaturation for the treatment of women with urinary incontinence. Cochrane Database Syst Rev. 2015 Mar 18;2015(3):CD010217. doi: 10.1002/14651858.CD010217.pub2. PMID 25785555
- [Result] Lordelo P, Vilas Boas A, Sodre D, Lemos A, Tozetto S, Brasil C. New concept for treating female stress urinary incontinence with radiofrequency. Int Braz J Urol. 2017 Sep-Oct;43(5):896-902. doi: 10.1590/S1677-5538.IBJU.2016.0621. PMID 28727373
- [Result] Imamura M, Abrams P, Bain C, Buckley B, Cardozo L, Cody J, Cook J, Eustice S, Glazener C, Grant A, Hay-Smith J, Hislop J, Jenkinson D, Kilonzo M, Nabi G, N'Dow J, Pickard R, Ternent L, Wallace S, Wardle J, Zhu S, Vale L. Systematic review and economic modelling of the effectiveness and cost-effectiveness of non-surgical treatments for women with stress urinary incontinence. Health Technol Assess. 2010 Aug;14(40):1-188, iii-iv. doi: 10.3310/hta14400. PMID 20738930
- [Result] Radziminska A, Straczynska A, Weber-Rajek M, Styczynska H, Strojek K, Piekorz Z. The impact of pelvic floor muscle training on the quality of life of women with urinary incontinence: a systematic literature review. Clin Interv Aging. 2018 May 17;13:957-965. doi: 10.2147/CIA.S160057. eCollection 2018. PMID 29844662
- [Result] Soave I, Scarani S, Mallozzi M, Nobili F, Marci R, Caserta D. Pelvic floor muscle training for prevention and treatment of urinary incontinence during pregnancy and after childbirth and its effect on urinary system and supportive structures assessed by objective measurement techniques. Arch Gynecol Obstet. 2019 Mar;299(3):609-623. doi: 10.1007/s00404-018-5036-6. Epub 2019 Jan 16. PMID 30649605
- [Result] Dumoulin C, Cacciari LP, Hay-Smith EJC. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005654. doi: 10.1002/14651858.CD005654.pub4. PMID 30288727
- [Result] Dumoulin C, Hay-Smith J, Frawley H, McClurg D, Alewijnse D, Bo K, Burgio K, Chen SY, Chiarelli P, Dean S, Hagen S, Herbert J, Mahfooza A, Mair F, Stark D, Van Kampen M; International Continence Society. 2014 consensus statement on improving pelvic floor muscle training adherence: International Continence Society 2011 State-of-the-Science Seminar. Neurourol Urodyn. 2015 Sep;34(7):600-5. doi: 10.1002/nau.22796. Epub 2015 May 21. PMID 25998603
- [Result] Sigurdardottir T, Steingrimsdottir T, Geirsson RT, Halldorsson TI, Aspelund T, Bo K. Can postpartum pelvic floor muscle training reduce urinary and anal incontinence?: An assessor-blinded randomized controlled trial. Am J Obstet Gynecol. 2020 Mar;222(3):247.e1-247.e8. doi: 10.1016/j.ajog.2019.09.011. Epub 2019 Sep 14. PMID 31526791
- [Result] Garcia-Sanchez E, Avila-Gandia V, Lopez-Roman J, Martinez-Rodriguez A, Rubio-Arias JA. What Pelvic Floor Muscle Training Load is Optimal in Minimizing Urine Loss in Women with Stress Urinary Incontinence? A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2019 Nov 8;16(22):4358. doi: 10.3390/ijerph16224358. PMID 31717291
- [Result] Hirakawa T, Suzuki S, Kato K, Gotoh M, Yoshikawa Y. Randomized controlled trial of pelvic floor muscle training with or without biofeedback for urinary incontinence. Int Urogynecol J. 2013 Aug;24(8):1347-54. doi: 10.1007/s00192-012-2012-8. Epub 2013 Jan 11. PMID 23306768
- [Result] Smith AL, Wein AJ. Urinary incontinence: pharmacotherapy options. Ann Med. 2011;43(6):461-76. doi: 10.3109/07853890.2011.564203. Epub 2011 Jun 3. PMID 21639723
- [Result] Tsakiris P, Oelke M, Michel MC. Drug-induced urinary incontinence. Drugs Aging. 2008;25(7):541-9. doi: 10.2165/00002512-200825070-00001. PMID 18582143
- [Result] Giarenis I, Cardozo L. Managing urinary incontinence: what works? Climacteric. 2014 Dec;17 Suppl 2:26-33. doi: 10.3109/13697137.2014.947256. Epub 2014 Sep 6. PMID 25196507
- [Result] Ben Ami N, Dar G. What is the most effective verbal instruction for correctly contracting the pelvic floor muscles? Neurourol Urodyn. 2018 Nov;37(8):2904-2910. doi: 10.1002/nau.23810. Epub 2018 Aug 28. PMID 30152550
- [Result] Messelink B, Benson T, Berghmans B, Bo K, Corcos J, Fowler C, Laycock J, Lim PH, van Lunsen R, a Nijeholt GL, Pemberton J, Wang A, Watier A, Van Kerrebroeck P. Standardization of terminology of pelvic floor muscle function and dysfunction: report from the pelvic floor clinical assessment group of the International Continence Society. Neurourol Urodyn. 2005;24(4):374-80. doi: 10.1002/nau.20144. No abstract available. PMID 15977259
- [Result] Leibaschoff G, Izasa PG, Cardona JL, Miklos JR, Moore RD. Transcutaneous Temperature Controlled Radiofrequency (TTCRF) for the Treatment of Menopausal Vaginal/Genitourinary Symptoms. Surg Technol Int. 2016 Oct 26;29:149-159. PMID 27608749
- See also: Guy AW, Lehmann JF, Stonebridge JB (1974) Therapeutic application of electromagnetic power. Proc IEEE, 62, 65-75. — http://zoryglaser.com/wp-content/uploads/2020/05/THERAPEUTIC-APPLICATIONS-OF-ELECTROMAGNETIC-POWER.pdf
- See also: Rodríguez-Mansilla, J., González Sánchez, B., de Toro García, A. and González-López-Arza, M. (2013). Eficacia de la hipertermia como tratamiento en las tendinopatías. Rehabilitación, 47(3), pp.179-185. — http://www.elsevier.es/en-revista-rehabilitacion-120-articulo-eficacia-hipertermia-como-tratamiento-las-S0048712013000170